CLINICAL TRIAL: NCT03631862
Title: A Randomized Controlled Clinical Trial of Apatinib Combined With CHOP Regimen in the Treatment of Newly Diagnosed Peripheral T-cell Lymphoma
Brief Title: Treatment of Newly Diagnosed Peripheral T-cell Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital, Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx2018-5
Record Dates: First submitted 2018-08-12; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Newly Diagnosed Peripheral T-cell Lymphoma
Keywords: peripheral T-cell lymphoma; Apatinib; targeted therapy; RR; PFS
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — apatinib; VAP-cyclo protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib combined with CHOP regimen (Experimental): Apatinib: 250mg/d d1-21 po CHOP regimen(Cyclophosphamide,Vincristine,Epirubicin,Prednisone) ： Cyclophosphamide 750mg/d,ivgtt, d1;Vincristine,1.4g/m2,ivgtt, d1;Epirubicin,60mg/m2,ivgtt,d1;Prednisone 60mg/m2,po, d1-5
  Interventions: Drug: Apatinib; Drug: CHOP Regimen
- CHOP regimen (Experimental): CHOP regimen(Cyclophosphamide,Vincristine,Epirubicin,Prednisone) ： Cyclophosphamide 750mg/d,ivgtt, d1;Vincristine,1.4g/m2,ivgtt, d1;Epirubicin,60mg/m2,ivgtt,d1;Prednisone 60mg/m2,po, d1-5
  Interventions: Drug: CHOP Regimen

INTERVENTIONS:
Drug: Apatinib — Apatinib is an orally administrated small molecule receptor tyrosine kinase inhibitor selectively targeting VEGFR-2, showing anti-tumor activity across a broad range of advanced cancers.
  Other Names: Apatinib mesylate
  Arms: Apatinib combined with CHOP regimen
Drug: CHOP Regimen — CHOP regimen(Cyclophosphamide,Vindesine,Epirubicin,Prednisone)
  Other Names: CHOP

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Apatinib Combined With CHOP Regimen(cyclophosphamide, vincristine, epirubicin, prednisone in the treatment of newly diagnosed peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
Patients with peripheral T-cell lymphoma usually have a bad prognosis. These patients cannot be treated successfully with the conventional CHOP regimen. Apatinib is a small-molecule multitargeted tyrosine kinase inhibitor. The investigators have been proceeding this trial to evaluate the efficacy and safety of the Apatinib Combined With CHOP Regimen(cyclophosphamide, vincristine, epirubicin, prednisone in the treatment of newly diagnosed peripheral T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Age range 14-70 years old; ECOG performance status 0-2.
* Estimated survival time > 6 months.
* Histological confirmed Peripherial T-cell lymphoma.
* Have taken no treatment.
* None of chemotherapy contraindication: hemoglobin ≥ 90 g/dl, neutrophil ≥ 1.5×109/L, platelet ≥ 100×109/L, ALT and AST ≤ 2×ULN, serum bilirubin ≤ 1.5×ULN, serum creatine ≤ 1.5×upper limitation of normal (ULN), Serum Albumin ≥ 30g/L, serum plasminogen is normal.
* At least one measurable lesion.
* None of other serious diseases, cardiopulmonary function is normal.
* Pregnancy test of women at reproductive age must be negative.
* Patients could be followed up.
* None of other relative treatments including the traditional Chinese medicine, immunotherapy, biotherapy except anti-bone metastasis therapy and other symptomatic treatments.
* Volunteers who signed informed consent.

Exclusion Criteria:

* Patients with contraindications (active bleeding, ulcers, intestinal perforation, intestinal obstruction, 30 days after major surgery, hypertension uncontrollable drugs, grade III-IV cardiac insufficiency, severe liver and kidney dysfunction);
* Abnormal coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), with bleeding tendency or undergoing thrombolysis or anticoagulant therapy；
* Urine routine indicates urinary protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0 g;
* Disagreement on blood sample collection.
* Patients allergic of any of drug in this regimen or with metabolic disorder.
* Pregnant or lactating women.
* Serious medical illness likely to interfere with participation.
* Serious infection.
* Primitive or secondary tumors of central nervous system.
* Chemotherapy or radiotherapy contraindication.
* The evidence of CNS metastasis.
* History of peripheral nervous disorder or dysphrenia.
* Patients participating in other clinical trials.
* Patients taking other antitumor drugs.
* Patients estimated to be unsuitable by investigator.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | up to end of follow-up-phase (approximately 24 months)
  Progression-free survival
RR | every 6 weeks, up to completion of treatment (approximately 18 weeks)
  Response Rate

SECONDARY OUTCOMES:
OS | up to the date of death (approximately 5 years)
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhi Zhang, Pro,Dr, Principal Investigator — China, Henan Oncology Department of The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Oncology Department of The First Affilliated Hospital of Zhengzhou University, Zhengzhou, Henan, China